CLINICAL TRIAL: NCT01506492
Title: Managing Cancer and Living Meaningfully (CALM): A Randomized Controlled Trial of a Psychotherapeutic Intervention for Patients With Metastatic Cancer
Brief Title: Managing Cancer and Living Meaningfully (CALM): A Study to Evaluate the Effectiveness of a Psychological Intervention for Cancer Patients
Acronym: CALM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 09-0855-C; CIHR (Other Grant/Funding Number: CIHR-MOP106473)
Record Dates: First submitted 2012-01-04; First posted 2012-01-10 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Depression
Keywords: Randomized controlled trial; Depression; Cancer; Psychotherapy; Quality of life
MeSH Terms: conditions — Depression; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention): Usual care includes routine screening for depression and other distress in oncology outpatient clinics, communication of screening information to the medical treatment team, and referral as needed.
- CALM (Experimental): Patients assigned to the intervention arm will receive 3-6 CALM therapy sessions over 3-6 months delivered by a trained therapist at our center.
  Interventions: Behavioral: CALM

INTERVENTIONS:
Behavioral: CALM — Patients assigned to the intervention arm will receive 3-6 CALM therapy sessions over 3-6 months delivered by a trained therapist at our center.
  Arms: CALM

SUMMARY:
The purpose of this study is to test the effectiveness of a brief manualized individual psychotherapy, called Managing Cancer and Living Meaningfully (CALM), to reduce distress and promote psychological well-being in patients with various types of cancer, including metastatic disease.

DETAILED DESCRIPTION:
We have developed and pilot-tested a brief manualized individual psychotherapy, called Managing Cancer and Living Meaningfully (CALM), to reduce distress in patients with various types of cancer, including metastatic disease. We propose to conduct a two-arm randomized controlled trial (RCT) to test the effectiveness of CALM against usual care (UC) for the reduction of distress in patients with various types of cancer, including metastatic disease. Usual care at our center includes routine screening for depression and other distress in oncology outpatient clinics, communication of screening information to the medical treatment team, and referral as needed for non-standardized, and primarily instrumental, psychosocial care and psychiatric assessment and treatment.

The design will be an unblinded RCT consisting of two conditions (CALM and UC), with a baseline assessment and follow-ups at three and six months. The trial will take place in Princess Margaret Cancer Centre, University Health Network, a comprehensive cancer center in Toronto, Canada. Participants will be outpatients with various types of cancer, including metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Fluency in English
* Confirmed diagnosis of stage III or IV lung cancer; any stage of pancreatic cancer, unresectable cholangiocarcinoma, unresectable liver cancer, unresectable ampullary/peri-ampullary cancer, or other stage IV (metastatic) gastrointestinal cancer; stage III or IV ovarian and fallopian tube cancers, or other stage IV gynecological cancers; and stage IV breast, genitourinary, sarcoma, melanoma or endocrine cancers (all with expected survival of 12-18 months)

Exclusion Criteria:

* Major communication difficulties (including language barriers)
* Inability to commit to the required 3-6 psychotherapy sessions
* Cognitive impairment indicated in the medical record, or by the attending oncologist, or as indicated by a score < 20 on the Short Orientation-Memory-Concentration test, unless deemed suitable at the recruiter's discretion
* Actively seeing a psychiatrist or psychologist in the Department of Supportive Care (formerly the Department of Psychosocial Oncology and Palliative Care) at Princess Margaret Cancer Centre at the time of study approach

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2012-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | 6-months
  A reliable and valid 9-item measure of depression that has been used widely with advanced cancer patients.

SECONDARY OUTCOMES:
Structured Clinical Interview for DSM Disorders (SCID)-Research Version | 6-months
  A semi-structured interview that allows researchers to make clinical diagnoses according to DSM criteria. Portions of the Mood Disorders and Optional Disorders modules will be administered: major depressive episode and minor depressive disorder.
Generalized Anxiety Disorders-7 (GAD-7) | 6-months
  A widely used and validated 7-item self-report measure designed to screen and assess the severity of GAD symptoms.
Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being Scale (FACIT-Sp) | 6-months
  A 12-item self-report measure of spiritual well-being, assessing spiritual meaning and peace, and faith, that has been widely used in palliative care research.
Posttraumatic Growth Inventory (PTGI) | 6-months
  A 21-item self-report scale that measures positive psychological changes after trauma. It has been used as a measure of psychological growth in cancer and as an outcome measure for intervention studies.
Quality of Life at the End of Life-Cancer Scale (QUAL-EC) | 6-months
  A measure of quality of life in patient populations near the end of life.
Death and Dying Distress Scale (DADDS) | 6-months
  A recently developed, 15-item measure assessing death anxiety in patients with advanced cancer.
Demoralization Scale (DS) | 6-months
  A 24-item self-report measure that assesses one aspect of existential distress, which includes loss of meaning and purpose, disheartenment and helplessness.
Experiences in Close Relationships Inventory Modified Short Form Version (ECR-M-16) | 6-months
  A 16-item self-report measure of attachment security.
Couple Communication Scale (CCS) | 6-months
  A measure for participants who are married, common-law, or in a long-term relationship. This measure is concerned with an individual's feelings, beliefs, and attitudes about the communication in his/her relationship.
Clinical Evaluation Questionnaire (CEQ) | 6-months
  A 7-item measure evaluating the extent to which patients felt emotionally supported by the clinical services provided.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Rodin, MD, Principal Investigator — University Health Network, Toronto; Sarah Hales, MD, PhD, Principal Investigator — University Health Network, Toronto; Chris Lo, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Nissim R, Freeman E, Lo C, Zimmermann C, Gagliese L, Rydall A, Hales S, Rodin G. Managing Cancer and Living Meaningfully (CALM): a qualitative study of a brief individual psychotherapy for individuals with advanced cancer. Palliat Med. 2012 Jul;26(5):713-21. doi: 10.1177/0269216311425096. Epub 2011 Oct 31. PMID 22042225
- [Background] Krause S, Rydall A, Hales S, Rodin G, Lo C. Initial validation of the Death and Dying Distress Scale for the assessment of death anxiety in patients with advanced cancer. J Pain Symptom Manage. 2015 Jan;49(1):126-34. doi: 10.1016/j.jpainsymman.2014.04.012. Epub 2014 May 28. PMID 24878066
- [Background] Lo C, Hales S, Jung J, Chiu A, Panday T, Rydall A, Nissim R, Malfitano C, Petricone-Westwood D, Zimmermann C, Rodin G. Managing Cancer And Living Meaningfully (CALM): phase 2 trial of a brief individual psychotherapy for patients with advanced cancer. Palliat Med. 2014 Mar;28(3):234-42. doi: 10.1177/0269216313507757. Epub 2013 Oct 29. PMID 24170718
- [Background] Neel C, Lo C, Rydall A, Hales S, Rodin G. Determinants of death anxiety in patients with advanced cancer. BMJ Support Palliat Care. 2015 Dec;5(4):373-80. doi: 10.1136/bmjspcare-2012-000420. Epub 2013 Aug 22. PMID 24644177
- [Background] Lo C, Hales S, Rydall A, Panday T, Chiu A, Malfitano C, Jung J, Li M, Nissim R, Zimmermann C, Rodin G. Managing Cancer And Living Meaningfully: study protocol for a randomized controlled trial. Trials. 2015 Sep 3;16:391. doi: 10.1186/s13063-015-0811-1. PMID 26335704
- [Background] Lo C, Hales S, Zimmermann C, Gagliese L, Rydall A, Rodin G. Measuring death-related anxiety in advanced cancer: preliminary psychometrics of the Death and Dying Distress Scale. J Pediatr Hematol Oncol. 2011 Oct;33 Suppl 2:S140-5. doi: 10.1097/MPH.0b013e318230e1fd. PMID 21952572
- [Background] Hales S, Lo C, Rodin G. Managing Cancer And Living Meaningfully (CALM) Therapy (Chapter 62) In: Holland JC, Breitbart WS, Butow PN, Jacobsen PB, Loscalzo MJ, McCorkle R, editors. Psycho-Oncology. 3. New York: Oxford University Press; 2015. pp. 487-91.
- [Background] Lo C, Hales S, Chiu A, Panday T, Malfitano C, Jung J, Rydall A, Li M, Nissim R, Zimmermann C, Rodin G. Managing Cancer And Living Meaningfully (CALM): randomised feasibility trial in patients with advanced cancer. BMJ Support Palliat Care. 2019 Jun;9(2):209-218. doi: 10.1136/bmjspcare-2015-000866. Epub 2016 Jan 19. PMID 26787360
- [Background] Tong E, Deckert A, Gani N, Nissim R, Rydall A, Hales S, Rodin G, Lo C. The meaning of self-reported death anxiety in advanced cancer. Palliat Med. 2016 Sep;30(8):772-9. doi: 10.1177/0269216316628780. Epub 2016 Feb 8. PMID 26857360
- [Result] Rodin G, Lo C, Rydall A, Shnall J, Malfitano C, Chiu A, Panday T, Watt S, An E, Nissim R, Li M, Zimmermann C, Hales S. Managing Cancer and Living Meaningfully (CALM): A Randomized Controlled Trial of a Psychological Intervention for Patients With Advanced Cancer. J Clin Oncol. 2018 Aug 10;36(23):2422-2432. doi: 10.1200/JCO.2017.77.1097. Epub 2018 Jun 29. PMID 29958037
- [Derived] An E, Wennberg E, Nissim R, Lo C, Hales S, Rodin G. Death talk and relief of death-related distress in patients with advanced cancer. BMJ Support Palliat Care. 2020 Jun;10(2):e19. doi: 10.1136/bmjspcare-2016-001277. Epub 2017 Aug 2. PMID 28768681